CLINICAL TRIAL: NCT05940831
Title: Integration of a Patient-centered Mobile Health Intervention (Support-moms) Into Routine Antenatal Care to Improve Maternal Health in Uganda.
Brief Title: Mobile Health Intervention (Support-moms) in Antenatal Care to Improve Maternal Health in Uganda
Acronym: Support-Moms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mbarara University of Science and Technology (Other)
Collaborators: University of Alabama at Birmingham (Other); Harvard Medical School (HMS and HSDM) (Other); Massachusetts General Hospital (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: MUST-2023-06-29; 1R01HD111692-01 (NIH)
Record Dates: First submitted 2023-06-30; First posted 2023-07-11 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Maternal Health
Keywords: mhealth; antenatal care; social support; healthcare utilization

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Scheduled SMS-audio messages from the final messaging prototype (SM), messages, plus social supporter engagement through SMS (SS)
  Interventions: Behavioral: Support-Moms
- Control (Active Comparator): Routine care/ information giving
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Support-Moms — Scheduled SMS-audio messages from the final messaging prototype (SM), plus social supporter engagement through SMS (SS).
  Arms: Intervention
Behavioral: Control — Routine care/ information giving
  Arms: Control

SUMMARY:
High maternal mortality is a major public health problem in many settings. Because of low antenatal care (ANC) and skilled birth usage, Ugandan women and their children suffer from high maternal and perinatal mortality. The investigators developed a promising intervention (Support-Moms app) that shares targeted health information, and engages social support networks through scheduled reminders to help support pregnant women to utilize maternity services in rural Uganda. The investigators now propose to test and implement the Support-Moms intervention and hypothesize that Support-Moms will be feasible and cost-effective in improving utilization of available maternity care services, and ultimately reduce maternal and perinatal mortality.

DETAILED DESCRIPTION:
Antenatal care (ANC) and skilled births are mainstays of preventing maternal and perinatal morbidity and mortality. Despite expanded availability of skilled birth attendants and referral health systems, Ugandan women have low ANC use and skilled births, resulting in one of the highest maternal mortality ratios and perinatal mortality rates in the world. Mobile health (mHealth) interventions can support individuals to internalize risks, need, and benefits of health services with high intervention delivery success. Provision of multiple messaging approaches-such as scheduled SMS, telephone voice messages and social support engagement-can empower individuals to seek and access care, and improve health outcomes. However, despite successes in pilot studies, there is little data on effectiveness, appropriateness, feasibility, fidelity and incremental costs needed to adopt, or scale up such strategies in sub-Saharan Africa, where the public health impact of such interventions is likely to be the greatest.

As part of a K43 career development award (PI Atukunda), the investigators used behavioral frameworks to develop a user-centered mHealth-based, audio-SMS messaging application to support pregnant individuals to use maternity care services in rural Uganda (Support-Moms app). The app shared health-related information and engaged social support networks via scheduled SMS/audio reminders and upcoming ANC appointment notifications. In a randomized 3-arm pilot study (n=120) comparing standard of care (SOC), scheduled messaging (SM), and scheduled messaging plus social supporter engagement (SS), the investigators observed high intervention uptake, acceptability, and feasibility. All women whose social supporters were engaged on the app attended ≥4 ANC visits, compared to 83% and 50% of women receiving only messages and SOC, respectively. Nearly all women in the SS arm (98%) had a skilled delivery compared to 78% and 70% in SM and SOC groups, respectively. The investigators now propose a type 1 hybrid implementation-effectiveness trial to evaluate and implement the Support-Moms intervention into routine care. The investigators will test the effectiveness of the intervention in a randomized controlled trial (N=824); the primary outcome will be the proportion of healthcare provider-led skilled births (Aim 1). The investigators will apply Proctor's implementation outcomes framework to evaluate implementation, service and client outcomes, and conduct in-depth interviews with users and key stakeholders to contextualize/clarify these outcomes, and explore implementation strategies for future scale-up using the Consolidated Framework for Implementation Research (CFIR) (Aim 2). They will assess costs and cost-effectiveness of implementing Support-Moms into routine care (Aim 3). The investigators hypothesize that Support-Moms will be an effective and cost-effective strategy to improve maternity service utilization.

ELIGIBILITY:
Inclusion Criteria:

Individuals who:

* are in the first trimester of pregnancy who have not yet presented for ANC
* reside in the catchment area of a study HC
* are emancipated minors and adults aged ≥ 18 years
* report access to a cell phone with reception in their home
* are able to identify at least two social supporters living within the study districts
* are able to provide consent.
* are from participants' existing social support network, with whom they have had stable, long-term relationships

Exclusion Criteria:

Participants will be excluded from the study if they:

* do not own a cell phone for personal use with reported reliable reception
* are unable to use SMS or unwilling to receive SMS notifications

Potential social supporters will be excluded from the study if they:

* are under 18 years of age
* do not own a cell phone for personal use with reported reliable reception
* are unable to use SMS or unwilling to receive SMS notifications
* have not had stable, long-term relationships with the participants
* are not aware that the study participant is pregnant

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1680 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2028-02-29 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
Healthcare provider (HCP)-led skilled births | 15 months
  Proportion of individuals delivering with the help of a healthcare provider (HCP)

SECONDARY OUTCOMES:
Maternal, implementation, service and client outcomes | 15 months
  Proportion of individuals who report the following outcomes: a) number of ANC visits, b) institution-based delivery, c) social support d) mode of infant delivery, e) all deaths (maternal, fetal, newborn), f) preterm birth, g) birth weight, h) breastfeeding, i) completion of post-natal care, j) complications of pregnancy and childbirth (e.g obstructed labor, ruptured uterus, need for neonatal or maternal resuscitation/ assisted ventilation, severe preeclampsia/ eclampsia, postpartum hemorrhage (PPH), maternal/newborn sepsis, and other infections); and implementation, service and client outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Esther C. Atukunda, PhD, Principal Investigator — Mbarara University of Science and Technology
Locations (2):
- Uganda (2):
  - Mbarara city, Mbarara
  - Mbarara district, Mbarara

IPD SHARING:
Plan to Share IPD: Yes
Sufficient patient/participant and facility data from this project will be preserved and shared to validate and replicate research findings described in our Aims. We are aware of the policies and guidelines established by NIH for Data Management and Strategy, and we intend to release and share all final research data and materials from this NIH-supported study for use by other researchers in a timely manner. We will endeavour to make accessible, the research tools to other researchers under reasonable terms and conditions promoting free competition and enterprise and reflecting dual obligations of disseminating unique research resources. The privacy and confidentiality of participants will be safeguarded at all time.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Ongoing
Access Criteria: Password protected through RedCap

REFERENCES:
- [Derived] Atukunda EC, Mugyenyi GR, Haberer JE, Siedner MJ, Musiimenta A, Najjuma JN, Obua C, Matthews LT. Integration of a Patient-Centered mHealth Intervention (Support-Moms) Into Routine Antenatal Care to Improve Maternal Health Among Pregnant Women in Southwestern Uganda: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Mar 19;14:e67049. doi: 10.2196/67049. PMID 40105879